CLINICAL TRIAL: NCT02559908
Title: A Multicenter, Single-blind, Randomized, Controlled Study of the Safety and Effectiveness of VYC-25L Hyaluronic Acid Injectable Gel for Restoration and Creation of Facial Volume in the Chin and Jaw
Brief Title: A Study of Hyaluronic Acid Injectable Gel (VYC-25L) for Restoration and Creation of Facial Volume in the Chin and Jaw
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V25L-001
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Chin Retrusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group_VYC-25L (Experimental): VYC-25L injection into the chin and/or jaw areas on Day 1, volume determined by the investigator (up to 4.0 mLs) and repeat treatment if applicable
  Interventions: Device: Hyaluronic Acid Injectable Gel
- Control Group_No treatment then VYC-25L (Other): No treatment for 3 months followed by VYC-25L injection into the chin and/or jaw areas, volume determined by the investigator (up to 4.0 mLs) and repeat treatment if applicable.
  Interventions: Device: Hyaluronic Acid Injectable Gel

INTERVENTIONS:
Device: Hyaluronic Acid Injectable Gel — Hyaluronic Acid Injectable Gel (VYC-25L) injection into the chin and/or jaw areas (up to 4.0 mLs).

SUMMARY:
This study will evaluate the safety and performance of VYC-25L hyaluronic acid injectable gel for the restoration and creation of facial volume in participants seeking to increase projection of the chin and/or jaw.

ELIGIBILITY:
Inclusion Criteria:

-Has chin retrusion.

Exclusion Criteria:

* Has ever received or is planning to receive permanent facial implants during the study.
* Has tattoos, piercings, facial hair or scars that would interfere with visual assessments of the chin or jaw.
* Has dentures or any device covering part of the palate or plans to undergo any dental procedure other than prophylaxis during the study.
* Has undergone semipermanent dermal filler treatment to the chin or jaw within 36 months or is planning treatment during the study.
* Has undergone any surgery of the chin or jaw area within 24 months or a planned surgery during the study.
* Has undergone mesotherapy, cosmetic resurfacing, or botulinum toxin injections within 6 months or a planned treatment during the study.
* Has experienced trauma to the chin and jaw area within 6 months.
* Has been previously diagnosed with streptococcal disease.
* Has a history of anaphylaxis or allergy to lidocaine, hyaluronic acid or streptococcal protein.
* Has porphyria or untreated epilepsy.
* Has active autoimmune disease.
* Has current cutaneous or mucosal inflammatory or infectious processes, abscess, an unhealed wound, or a cancerous or pre-cancerous lesion.
* Is on a concurrent regimen of lidocaine or structurally-related local anesthetics or is on a concurrent regimen of drugs that reduce or inhibit hepatic metabolism.
* Has impaired cardiac conduction, severely impaired hepatic function, or severe renal dysfunction.
* Is on an ongoing regimen of anti-coagulation therapy.
* Is on an ongoing regimen of medications (eg, aspirin, ibuprofen) or other substances known to increase coagulation time (eg, herbal supplements with garlic or gingko biloba) within the past 10 days.
* Has begun using any over-the-counter or prescription oral or topical, anti-wrinkle products below the subnasale within 30 days before enrollment or is planning to begin using such products during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-02-26 (Actual); Primary Completion 2016-02-12 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Glabella-Subnasale-Pogonion (G-Sn-Pog) Angle | Baseline, Month 3

SECONDARY OUTCOMES:
Percentage of Responders based on the Investigator's Assessment of Improvement in the Chin and Jaw Area using the 5-point Global Aesthetic Improvement Scale (GAIS) | Month 3
Percentage of Responders based on the Participant's Assessment of Improvement in the Chin and Jaw Area using the 5-point GAIS | Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Smita Chawla, Study Director — Allergan, plc
Locations (10):
- France (2):
  - Cabinet medical Solferino, Paris
  - Centre de Chirurgie Esthetique, Toulouse
- Germany (6):
  - Hautzentrum Altenbochum - RuhrDERM Gemeinschaftspraxis Dr. med. Ardabili - Dr. med. Niesmann, Bochum
  - Dermatolgie Köln am Rhein, Cologne
  - Rosenpark Research Geschäftsbereich der Rosenparkklinik GmbH, Darmstadt
  - Rotes Kreuz Krankenhaus Kassel Gemeinnützige GmbH Klinik für Plastische, Rekonstruktive und Ästhetische Chirurgie, Kassel
  - Praxisgemeinschaft Theatiner46 Dres. Ogilvie und Dr. Bernd Schuster, Munich
  - Dermatogische Privatpraxis CentroDerm GmbH, Wuppertal
- Netherlands (2):
  - Kliniek Dokter Frodo Gaymans, Amsterdam
  - Joost Kroon Cosmetische Kliniek, Amsterdam

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com